CLINICAL TRIAL: NCT01294540
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Oral Doses of E2609 in Healthy Subjects and an Elderly Cohort
Brief Title: Evaluation of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E2609 in Healthy Subjects and an Elderly Cohort
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2609-A001-001
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: 1 (Experimental)
  Interventions: Drug: Drug: E2609
- Placebo Comparator: 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drug: E2609 — E2609 orally at varying ascending doses
  Arms: Experimental: 1
Drug: Placebo — Matching Placebo
  Arms: Placebo Comparator: 2

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of E2609 when administered as single doses to healthy adult volunteers and healthy elderly subjects. The study will consist of 2 parts:(1) a single dose in healthy adult volunteers, at doses up to 800 mg or the maximum dose that can be tolerated, (2) a single dose of 50 mg in healthy elderly volunteers.

DETAILED DESCRIPTION:
The study will consist of 2 parts: (1) a single dose in healthy adult volunteers, at doses up to 100 mg or the maximum dose that can be tolerated, (2) a single dose of 25 mg or lower in healthy elderly volunteers.

ELIGIBILITY:
Inclusion:

* Healthy males and females
* Aged 30 to 55 years, inclusive (Cohorts 1 through 5); aged 65 to 85 years, inclusive (Cohort 6)
* Body mass index (BMI) of 18 to 32kg/m^2 at Screening
* Additional inclusion criteria for Cohort 6 (healthy elderly subjects)

Exclusion

* Females of child-bearing potential
* Personal or family history of neurological abnormalities
* Any clinical abnormality of the electrocardiogram (ECG)at Screening and check-in
* A family history of cardiac abnormalities
* Thyroid abnormalities

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as evidenced by the number of subjects with adverse events | 38 days

SECONDARY OUTCOMES:
To assess the pharmacokinetics (PK) of E2609 in plasma and urine following administration of single oral doses | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yen, Principal Investigator — Glendale Adventist Medical Center, Glendale, California
Locations (1):
- Glendale Adventist Medical Center, Glendale, California, United States